CLINICAL TRIAL: NCT04005989
Title: Adipose Stromal Cells Injection in the Myocardium for Induction of Revascularization
Acronym: ADMIRE
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to logistic issues during COVID-19 pandemic
Sponsor: Hospital do Coracao (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADMIRE
Record Dates: First submitted 2019-06-13; First posted 2019-07-02 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2021-07

CONDITIONS: Ischemic Heart Disease; Myocardial Ischemia; Coronary Artery Disease
Keywords: STROMAL CELLS; ADIPOSE STROMAL CELLS; REVASCULARIZATION; MYOCARDIUM REVASCULARIZATION; CARDIAC SURGERY; CORONARY ARTERY DISEASE
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: It is a randomized, prospective, double-blind, placebo-controlled clinical study.
  Eligible patients will be randomly divided into 4 groups (one control group and 3 active treatment groups): 10 PATIENTS EACH ARM Control Group - saline injection Low dose group (BD) - hASC injection (1x106 / kg body weight) Intermediate dose group (DI) - injection of hASC (2x106 / kg body weight) High dose group (AD) - hASC injection (4x106 / kg body weight)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: DOUBLE BLIND
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PLACEBO GROUP (Placebo Comparator): injection of saline solution
  Interventions: Biological: Stromal Cells Injection
- Low dose group (Active Comparator): hASC injection (1x10e6 / kg body weight)
  Interventions: Biological: Stromal Cells Injection
- Intermediate Dose (Active Comparator): injection of hASC (2x10e6 / kg of body weight)
  Interventions: Biological: Stromal Cells Injection
- High dose group (Active Comparator): injection of hASC (4x10e6 / kg body weight)
  Interventions: Biological: Stromal Cells Injection

INTERVENTIONS:
Biological: Stromal Cells Injection — Adipose stromal cell

SUMMARY:
Treatment of ischemic myocardium has been the subject of intense research in recent years and stem cell therapy is one of the great promises. The InCor laboratory has studied cells from different backgrounds as candidates for cell therapy in the context of myocardial infarction. Evidence in preclinical studies of the application of stromal (mesenchymal) adipose tissue (hASC) in the ischemic heart by both the InCor group (in the animal model in rodents and pigs) and others in the literature suggest relevant benefits on the decrease of deterioration post-infarction. More recently it has been demonstrated that it arises mainly from the formation of new vessels due to paracrine factors, which are secreted by the injected cells. There are currently no studies in Brazil in which the safety of injecting different doses of hASC cells into the heart has been particularly evaluated. Recently, two studies have demonstrated the clinical applicability of hASC in patients with peripheral ischemic disease and stroke.

Thus, the objective of this work will be to test the hypothesis that the implantation of autologous stromal cells derived from adipose tissue combined with myocardial revascularization surgery in patients with coronary artery disease

DETAILED DESCRIPTION:
To test the hypothesis that the implantation of adipose-derived autologous cells derived from adipose tissue (hASCs) combined with coronary artery bypass grafting in patients with coronary artery disease is safe and well tolerated, besides being able to promote regional perfusion increase in the injected segments.

ELIGIBILITY:
Inclusion Criteria:

* signing the Informed Consent Form (TCLE)
* the patient must be a patient with obstructive atherosclerotic coronary artery disease
* sex: both men and women are eligible-
* Age: between 18 and 80 years of age
* the patient should present clinical evidence (angina pectoris or angina equivalent) OR imaging (stress echocardiography, myocardial perfusion scintigraphy, cardiac magnetic resonance imaging) of myocardial ischemia, invasively stratified with coronary angiography
* the presence of myocardial ischemia should be confirmed by at least 2 (two) distinct diagnostic methods performed within one year of the patient's inclusion in the study
* the patient is a candidate for myocardial revascularization surgery but coronary obstructive lesions, in their entirety, are NOT amenable for surgical treatment in the opinion of the surgeon (main surgeon), depending on the anatomical type, extent or distal involvement of the lesions OR, even if they can be treated surgically as a whole, an unsatisfactory surgical outcome is anticipated in terms of functional gain (restoration of myocardial perfusion)

Exclusion Criteria:

do not meet ALL criteria for inclusion

* have a concomitant severe disease, at an advanced stage, or with an unquestionable shortening of life expectancy (<1 year), or that prevents complementary examinations and / or attendance at follow-up visits
* have a confirmed diagnosis, previous history and / or past treatment of neoplasia, of any location and staging, in the last 5 years
* being in clinical treatment or awaiting surgical treatment of neoplasia, any location and staging
* present, during the outpatient investigation, unequivocal findings of neoplasia
* have symptoms attributable exclusively to left ventricular dysfunction, although of ischemic etiology, without the evidence of current myocardial ischemia, by at least two (2) methods of evaluation
* presented severe left ventricular dysfunction as defined by transthoracic echocardiography due to the finding of a left ventricular ejection fraction <0.25 (Simpson's method)
* have a history or current diagnosis of severe ventricular arrhythmias such as sustained ventricular tachycardia unless an automatic cardioverter-defibrillator has been implanted previously
* Concurrent heart diseases of other etiologies (valvular, idiopathic, hypertensive, Chagasic, etc.).
* have a history of acute coronary syndrome (unstable angina or acute myocardial infarction) in the last 3 months
* present chronic renal failure in dialysis treatment
* have participated in other cell therapy studies in the past 2 years
* Pregnant women
* patients diagnosed with acquired immunodeficiency syndrome (AIDS)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular Death | 12 months
  Death due to stroke, myocardial infarction or other cardiovascular causes
Unstable angina | 12 months
  Occurence of angina requiring hospitalization
Acute myocardial infarction | 12 months after procedure
  Occurence of acute myocardial infarction (with or without ST segment elevation)
Unplanned myocardial revascularization surgery | 12 months
  Need for urgent surgical myocardial revascularization
Unplanned myocardial revascularization through angioplasty | 12 months
  Need for urgent non-surgical myocardial revascularization

SECONDARY OUTCOMES:
All cause mortality | 12 months
Stroke | 12 months
Cardiogenic shock | 12 months
Occurence of complex ventricular arrhythmia | 12 months
New onset atrial fibrilation | 12 months
Occurence of acute pulmonary edema | 12 months
Pulmonary embolism | 12 months
Acute respiratory failure of any cause | 12 months
Septic shock | 12 months
  Disseminated infection requiring vasopressors
New onset cancer | 12 month
  Diagnosis of any cancer at any stage during study period